CLINICAL TRIAL: NCT04312464
Title: Retrospective Study of Myocardial Damage in COVID-19
Brief Title: Myocardial Damage in COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: MD-COVID-19
Record Dates: First submitted 2020-03-04; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: COVID-19; Cardiovascular Diseases
Keywords: COVID-19; myocardial injury
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discharged group: The individual which is defined as patient discharged from hospital
  Interventions: Other: non
- Dead group: The individual which is defined as patient with all-cause death
  Interventions: Other: non

INTERVENTIONS:
Other: non — no intervention

SUMMARY:
This study aims to investigate the clinical characteristics, the incidence of myocardial injury, and the influence of myocardial injury on the prognosis in COVID-19 patients. There is no additional examination and treatment for this project.

DETAILED DESCRIPTION:
The epidemic of the COVID-19 has expanded from Wuhan through out China, and is being exported to a growing number of countries. Recently, investigators have revealed that acute myocardial injury is existed in 7.2% patients with COVID-19, and this proportion in patients admitted to the ICU (22.2%) is higher than patients not treated in the ICU (2.0%). Thus, cardiac troponin I (cTNI), the biomarker of cardiac injury, might be a clinical predictor of COVID-19 patient outcomes. This study aims to investigate the clinical characteristics, the incidence of myocardial injury, and the influence of myocardial injury on the prognosis in COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years. (2) Laboratory (RT-PCR) confirmed infection with SARS-CoV-2. (3) Lung involvement confirmed with chest imaging.

Exclusion Criteria:

* No cTnI test on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The laboratory-confirmed patients with confirmed COVID-19 admitted to headquarters, west campus and cancer center of Union Hospital, Tongji Medical College, Huazhong University of science and technology, from January 1st to March 15th, 2020
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-15 (Estimated); Study Completion 2020-03-18 (Estimated)

PRIMARY OUTCOMES:
The myocardial injury incidence | 75 days
  The myocardial injury incidence of COVID-19 patients
The risk factors analysis for the death | 75 days
  The risk factors analysis for the death of COVID-19 patients

SECONDARY OUTCOMES:
Clinical characteristics | 75 days
  The clinical characteristics description of COVID-19 patients
Clinical course | 75 days
  The clinical course description of COVID-19 patients
Cardiovascular comorbidity | 75 days
  The clinical characteristics and prognosis analysis in different cardiovascular comorbidity of COVID-19 patients
Analysis of causes of death | 75 days
  Analysis of causes of death in COVID-19 patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China